CLINICAL TRIAL: NCT02163161
Title: A Phase 1, Open Label, Single Dose 3 Way Crossover Study to Evaluate the Bioavailability of a Solid Dose Formulation of PF 04965842 Relative to a Suspension Formulation Under Fasting Conditions and the Effect of Food on the Bioavailability of the Solid Dosage Formulation of Pf 04965842 in Healthy Subjects
Brief Title: AStudy to Evaluate the Bioavailability of PF 04965842 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7451004
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Phase I; Open Label; Single dose; Crossover; Bioavailability; Fasting; Fed; PF-04965842; Healthy
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: PF-04965842
- Treatment B (Experimental)
  Interventions: Drug: PF-04965842
- Treatment C (Experimental)
  Interventions: Drug: PF- 04965842

INTERVENTIONS:
Drug: PF-04965842 — Subjects will receive 4 x 100 mg PF 04965842 tablet under fasted conditions
  Arms: Treatment A
Drug: PF-04965842 — Subjects will receive 400 mg PF 04965842 oral suspension under fasted conditions
  Arms: Treatment B
Drug: PF- 04965842 — Subjects will receive 4 x 100 mg PF 04965842 tablet under fed conditions
  Arms: Treatment C

SUMMARY:
Phase 1, open label, single dose, 3 way crossover study to evaluate the bioavailability of a solid dose formulation of PF 04965842 relative to a suspension formulation under fasting conditions and the effect of food on the bioavailability of the solid dosage formulation of PF 04965842 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Subjects who received within 7 days prior to the first dose of study medication or are likely to receive during the study any moderate strong inhibitors of CYP3A4, eg, itraconazole, erythromycin, ketoconazole, protease inhibitors, verapamil, or diltiazem.
* Subjects who received within 28 days or are likely to receive during the study inducers of CYP3A4, eg rifampin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from Time Zero to infinity (AUC inf) | 15 days
Maximum Observed Plasma Concentration (Cmax) | 15 days
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 15 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 15 days
Plasma Decay Half-Life (t1/2) | 15 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451004&StudyName=AStudy%20to%20Evaluate%20the%20Bioavailability%20of%20%20PF%2004965842%20in%20Healthy%20Subjects%20